CLINICAL TRIAL: NCT04985435
Title: Better After CHoosing. Randomly Allocated or Patient Preference Based Treatment With Filgotinib or TNFi in Patients With Active Rheumatoid Arthritis (BACH)
Brief Title: Better After CHoosing. Randomly Allocated or Patient Preference Based Treatment With Filgotinib or TNFi in RA (BACH)
Acronym: BACH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: R.Bos (Other)
Collaborators: Galapagos NV (Industry); Frisius Medisch Centrum (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor-Investigator, R.Bos, principal (coordinating) investigator, Rheumatology Research Center Northern Netherlands
Organization: Rheumatology Research Center Northern Netherlands (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTPO 1111; NL76371.099.21 (Other: CCMO ABR number)
Record Dates: First submitted 2021-07-19; First posted 2021-08-02 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634; Pharmaceutical Preparations; Adalimumab; Etanercept

STUDY DESIGN:
Intervention Model Description: randomized open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Choice group (Active Comparator): 50 patients will be randomized to the choice group, they will view a neutral information video on anti TNF and Filgotinib and will be given the opportunity to choose between these two treatments
  Interventions: Drug: Filgotinib; Drug: Anti-Tumor Necrosis Factor Alpha Drug (Product); Behavioral: 50 patients will have a Free Choice between Filgotinib and anti TNF
- Randomization group anti TNF (Active Comparator): A total of 50 patients will be randomized to the randomization group: 25 of those will start treatment with antiTNF
  Interventions: Drug: Anti-Tumor Necrosis Factor Alpha Drug (Product)
- Randomization group Filgotinib (Active Comparator): A total of 50 patients will be randomized to the randomization group: 25 of those will start treatment with Filgotinib
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — 200 mg tablet once daily or 100 mg once daily
  Other Names: Jyseleca
  Arms: Choice group; Randomization group Filgotinib
Drug: Anti-Tumor Necrosis Factor Alpha Drug (Product) — Adalimumab subcutaneous injections 40 mg once every two weeks Etanercept subcutaneous injections 50 mg weekly
  Other Names: Adalimumab (Humira) Etanercept (Enbrel)
  Arms: Choice group; Randomization group anti TNF
Behavioral: 50 patients will have a Free Choice between Filgotinib and anti TNF — 50 patients will be given the opportunity to choose between either TNFi (etanercept 50 mg SC once a week or adalimumab 40 mg SC once every two weeks) or filgotinib, an oral JAKi, 200 mg once a day while another group of 50 patients will be randomized to the same treatment arms.
  Arms: Choice group

SUMMARY:
Despite their efficacy in the treatment of Rheumatoid Arthritis and their partial advantage over traditional bDMARDs ( biological Disease Modifying antirheumatic drugs), JAK inhibitors (JAKi or tsDMARDs) have not gained preference over Tumor Necrosis Factor inhibitors (TNFi) in guidelines or clinical practice. The biggest influence on recent guidelines has been the "Treat To Target" principle (T2T), in which Shared Decision Making (SDM) plays a key part. Patient preference has proven to be a large barrier in treatment adjustments (14- 37%) while patients showed better adherence and higher treatment satisfaction when engaged in Shared Decision Making. From survey studies it is suggested that patient preference and satisfaction will be in favour of oral JAK inhibitors over parenteral biologics.The investigators want to establish the treatment preference of patients with active RA and compare the treatment satisfaction of patients who are given the opportunity to choose between the JAKi filgotinib and TNFi, to the treatment satisfaction of patients who are randomized to the same treatment options.

In addition to higher treatment satisfaction and better adherence, the investigators expect to find an improvement in DAS28-, HAQ-, SQUASH- and WPAI-scores and also an improved activity and work productivity.

DETAILED DESCRIPTION:
Rationale: Despite their efficacy in the treatment of Rheumatoid Arthritis and their partial advantage over traditional bDMARDs, JAK inhibitors (JAKi or tsDMARDs) have not gained preference over Tumor Necrosis Factor inhibitors (TNFi) in guidelines or clinical practice. The biggest influence on recent guidelines has been the "Treat To Target" principle (T2T), in which Shared Decision Making (SDM) plays a key part. Patient preference has proven to be a large barrier in treatment adjustments (14- 37%) while patients showed better adherence and higher treatment satisfaction when engaged in Shared Decision Making. From survey studies it is suggested that patient preference and satisfaction will be in favour of oral JAK inhibitors over parenteral biologics. The investigators want to establish the treatment preference of patients with active RA and compare the treatment satisfaction of patients who are given the opportunity to choose between the JAKi filgotinib and TNFi, to the treatment satisfaction of patients who are randomized to the same treatment options.

In addition to higher treatment satisfaction and better adherence, the investigators expect to find an improvement in DAS28-, HAQ-, SQUASH- and WPAI-scores and also an improved activity and work productivity.

Objective:

* To evaluate the actual preference of patients when they decide themselves which mode of action they want to use for treatment of rheumatoid arthritis.
* To evaluate differences in treatment satisfaction between patients who can choose their therapy and those patients that are randomized for the same treatment options.
* To evaluate if adherence to therapy is increased when patients decide their own therapy.
* To evaluate the difference in improvement of disease activity by the Disease Activity Score (DAS28) and physical activity as measured by SQUASH questionnaire and fitness trackers.

Study design: This study is a multicenter, randomized, 24-week, open label trial

Study population and intervention:

Early, bDMARD naive RA patients, of whom a group of 50 patients will be given the opportunity to choose between either TNFi (etanercept 50 mg SC once a week or adalimumab 40 mg SC once every two weeks) or filgotinib, an oral JAKi, 200 mg once a day while another group of 50 patients will be randomized to the same treatment arms.

Main study parameters/endpoints: The two primary endpoints consist of:

* The proportion of subjects in the first subgroup choosing filgotinib therapy at baseline
* Treatment satisfaction of both subgroups at week 24 at a 5-point Likert scale for current medical treatment.

Burden and risks associated with participation, benefit and group relatedness: All medication is prescribed at the indicated dosages used in clinical care, according to international guidelines. Study burden and risks are similar to daily clinical care: In addition to daily clinical care one half of the participants has to make the treatment choice and all participants will fill in questionnaires, which will take about 15 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

Demographic and general characteristics:

* Adult male or female patients, at least 18 years of age.
* Able and willing to give written informed consent.
* Have sufficient knowledge of the Dutch language to be able to comply with the requirements of the study protocol.

Inclusion criteria:

* Diagnosis of adult-onset RA as defined by the 2010 ACR/ EULAR Rheumatoid arthritis classification criteria;
* Diagnosis of RA for ≥ three months;
* Are being treated ≥ three months with ≥ 1 csDMARD therapy;
* Have had an inadequate response or intolerance to at least 1 csDMARD;
* Have moderately to severely active RA to the discretion of the rheumatologist or defined as a DAS28 ≥ 3.2 at screening and baseline visits;
* Subjects must have been on a stable dose of csDMARD therapy (restricted to methotrexate, chloroquine, hydroxychloroquine, sulfasalazine, or leflunomide) for ≥ 4 weeks prior to the baseline visit.

Exclusion Criteria:

* Previous treatment with any biological DMARD or targeted synthetic DMARD/JAKi;
* Inflammatory rheumatic disease other than RA, except for secondary Sjögren's syndrome.
* Having a contraindication for either TNFi or filgotinib;
* Latent or active tuberculosis;
* Active or recurrent infections;
* History of any malignancy within 5 years except for successfully treated NMSC or localized carcinoma in situ of the cervix;
* ≥ 3x upper limit of normal ALT, AST;
* eGFR ≤ 30 ml/min;
* planned or actual pregnancy or planning to father a child.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects in the first subgroup choosing filgotinib therapy at baseline | Baseline data
  The proportion of subjects in the first subgroup choosing filgotinib therapy at baseline
Treatment satisfaction at week 24 | 24 weeks
  Treatment satisfaction of both subgroups at week 24 at a 5-point Likert scale for current medical treatment: Ranging from 1: very dissatisfied, 2: dissatisfied, 3: neither dissatisfied nor satisfied, 4: satisfied, 5: very satisfied.

SECONDARY OUTCOMES:
How patients rate being informed by the neutral information video | week 6 and week 24
  How patients rate being informed by the neutral information video on a Likert scale of agreement on being well informed, ranging from 1: strongly disagree, 2: disagree, 3: undecided, 4: agree, 5: strongly agree
How do patients in the treatment Choice group I rate being in control for their treatment decision. | week 6 and week 24
  How do patients in the treatment Choice group I rate being in control for their treatment decision.
Proportion of subjects who would choose filgotinib (again or otherwise) at 24-weeks if they were allowed to choose again. | week 24
  Proportion of subjects who would choose filgotinib (again or otherwise) at 24-weeks if they were allowed to choose again.
Proportion of patients who were not able to make a treatment decision. | baseline data
  Proportion of patients who were not able to make a treatment decision.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Bos, MD PhD, Principal Investigator — Rheumatology Research Center Northern Netherlands
Locations (1):
- Medical Center Leeuwarden MCL, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zak A, Corrigan C, Yu Z, Bitton A, Fraenkel L, Harrold L, Smolen JS, Solomon DH. Barriers to treatment adjustment within a treat to target strategy in rheumatoid arthritis: a secondary analysis of the TRACTION trial. Rheumatology (Oxford). 2018 Nov 1;57(11):1933-1937. doi: 10.1093/rheumatology/key179. PMID 29982720
- [Background] Schipper LG, Vermeer M, Kuper HH, Hoekstra MO, Haagsma CJ, Den Broeder AA, van Riel P, Fransen J, van de Laar MA. A tight control treatment strategy aiming for remission in early rheumatoid arthritis is more effective than usual care treatment in daily clinical practice: a study of two cohorts in the Dutch Rheumatoid Arthritis Monitoring registry. Ann Rheum Dis. 2012 Jun;71(6):845-50. doi: 10.1136/annrheumdis-2011-200274. Epub 2011 Dec 30. PMID 22210852
- [Background] Tymms K, Zochling J, Scott J, Bird P, Burnet S, de Jager J, Griffiths H, Nicholls D, Roberts L, Arnold M, Littlejohn G. Barriers to optimal disease control for rheumatoid arthritis patients with moderate and high disease activity. Arthritis Care Res (Hoboken). 2014 Feb;66(2):190-6. doi: 10.1002/acr.22108. PMID 23983001
- [Background] Lofland JH, Johnson PT, Ingham MP, Rosemas SC, White JC, Ellis L. Shared decision-making for biologic treatment of autoimmune disease: influence on adherence, persistence, satisfaction, and health care costs. Patient Prefer Adherence. 2017 May 18;11:947-958. doi: 10.2147/PPA.S133222. eCollection 2017. PMID 28572722
- [Background] Alten R, Kruger K, Rellecke J, Schiffner-Rohe J, Behmer O, Schiffhorst G, Nolting HD. Examining patient preferences in the treatment of rheumatoid arthritis using a discrete-choice approach. Patient Prefer Adherence. 2016 Nov 1;10:2217-2228. doi: 10.2147/PPA.S117774. eCollection 2016. PMID 27843301
- [Background] Schiffner-Rohe J, Alten R, Kruger K, Behmer OS, Schiffhorst G, Rellecke J, Nolting HD. Patient Preferences in the Choice of Disease Modifying Anti-Rheumatic Drugs. Value Health. 2014 Nov;17(7):A385. doi: 10.1016/j.jval.2014.08.2641. Epub 2014 Oct 26. No abstract available. PMID 27200872
- [Background] Taylor PC, Betteridge N, Brown TM, Woolcott J, Kivitz AJ, Zerbini C, Whalley D, Olayinka-Amao O, Chen C, Dahl P, Ponce de Leon D, Gruben D, Fallon L. Treatment Mode Preferences in Rheumatoid Arthritis: Moving Toward Shared Decision-Making. Patient Prefer Adherence. 2020 Jan 20;14:119-131. doi: 10.2147/PPA.S220714. eCollection 2020. PMID 32021123
- [Background] Goekoop-Ruiterman YP, de Vries-Bouwstra JK, Allaart CF, van Zeben D, Kerstens PJ, Hazes JM, Zwinderman AH, Ronday HK, Han KH, Westedt ML, Gerards AH, van Groenendael JH, Lems WF, van Krugten MV, Breedveld FC, Dijkmans BA. Clinical and radiographic outcomes of four different treatment strategies in patients with early rheumatoid arthritis (the BeSt study): a randomized, controlled trial. Arthritis Rheum. 2005 Nov;52(11):3381-90. doi: 10.1002/art.21405. PMID 16258899
- [Background] van Eijk IC, Nielen MM, van der Horst-Bruinsma I, Tijhuis GJ, Boers M, Dijkmans BA, van Schaardenburg D. Aggressive therapy in patients with early arthritis results in similar outcome compared with conventional care: the STREAM randomized trial. Rheumatology (Oxford). 2012 Apr;51(4):686-94. doi: 10.1093/rheumatology/ker355. Epub 2011 Dec 13. PMID 22166255
- [Background] Schipper LG, van Hulst LT, Grol R, van Riel PL, Hulscher ME, Fransen J. Meta-analysis of tight control strategies in rheumatoid arthritis: protocolized treatment has additional value with respect to the clinical outcome. Rheumatology (Oxford). 2010 Nov;49(11):2154-64. doi: 10.1093/rheumatology/keq195. Epub 2010 Jul 29. PMID 20671022
- [Background] Goekoop-Ruiterman YP, de Vries-Bouwstra JK, Kerstens PJ, Nielen MM, Vos K, van Schaardenburg D, Speyer I, Seys PE, Breedveld FC, Allaart CF, Dijkmans BA. DAS-driven therapy versus routine care in patients with recent-onset active rheumatoid arthritis. Ann Rheum Dis. 2010 Jan;69(1):65-9. doi: 10.1136/ard.2008.097683. PMID 19155234
- [Background] Smolen JS, Breedveld FC, Burmester GR, Bykerk V, Dougados M, Emery P, Kvien TK, Navarro-Compan MV, Oliver S, Schoels M, Scholte-Voshaar M, Stamm T, Stoffer M, Takeuchi T, Aletaha D, Andreu JL, Aringer M, Bergman M, Betteridge N, Bijlsma H, Burkhardt H, Cardiel M, Combe B, Durez P, Fonseca JE, Gibofsky A, Gomez-Reino JJ, Graninger W, Hannonen P, Haraoui B, Kouloumas M, Landewe R, Martin-Mola E, Nash P, Ostergaard M, Ostor A, Richards P, Sokka-Isler T, Thorne C, Tzioufas AG, van Vollenhoven R, de Wit M, van der Heijde D. Treating rheumatoid arthritis to target: 2014 update of the recommendations of an international task force. Ann Rheum Dis. 2016 Jan;75(1):3-15. doi: 10.1136/annrheumdis-2015-207524. Epub 2015 May 12. PMID 25969430
- [Background] Smolen JS, Landewe RBM, Bijlsma JWJ, Burmester GR, Dougados M, Kerschbaumer A, McInnes IB, Sepriano A, van Vollenhoven RF, de Wit M, Aletaha D, Aringer M, Askling J, Balsa A, Boers M, den Broeder AA, Buch MH, Buttgereit F, Caporali R, Cardiel MH, De Cock D, Codreanu C, Cutolo M, Edwards CJ, van Eijk-Hustings Y, Emery P, Finckh A, Gossec L, Gottenberg JE, Hetland ML, Huizinga TWJ, Koloumas M, Li Z, Mariette X, Muller-Ladner U, Mysler EF, da Silva JAP, Poor G, Pope JE, Rubbert-Roth A, Ruyssen-Witrand A, Saag KG, Strangfeld A, Takeuchi T, Voshaar M, Westhovens R, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2019 update. Ann Rheum Dis. 2020 Jun;79(6):685-699. doi: 10.1136/annrheumdis-2019-216655. Epub 2020 Jan 22. PMID 31969328
- [Background] Louder AM, Singh A, Saverno K, Cappelleri JC, Aten AJ, Koenig AS, Pasquale MK. Patient Preferences Regarding Rheumatoid Arthritis Therapies: A Conjoint Analysis. Am Health Drug Benefits. 2016 Apr;9(2):84-93. PMID 27182427
- [Background] Barton JL. Patient preferences and satisfaction in the treatment of rheumatoid arthritis with biologic therapy. Patient Prefer Adherence. 2009 Nov 29;3:335-44. doi: 10.2147/ppa.s5835. PMID 20016797
- [Background] Raghunath S, Hijjawi R, Hoon E, Shanahan EM, Goldblatt F. Qualitative assessment of medication adherence in patients with rheumatic diseases on biologic therapy. Clin Rheumatol. 2019 Oct;38(10):2699-2707. doi: 10.1007/s10067-019-04609-y. Epub 2019 Jun 6. PMID 31172365
- [Background] Stalpers J. Psychological Determinants of Subjective health. Doctoral dissertation, Nyenrode Business Universiteit, The Netherlands. Nyenrode Business Universiteit. Doctoral dissertation, Nyenrode Business Universiteit, The Netherlands 2009;.
- [Background] Nota I, Drossaert CH, Taal E, van de Laar MA. Arthritis patients' motives for (not) wanting to be involved in medical decision-making and the factors that hinder or promote patient involvement. Clin Rheumatol. 2016 May;35(5):1225-35. doi: 10.1007/s10067-014-2820-y. Epub 2014 Nov 14. PMID 25392118
- [Background] Schildmann J, Grunke M, Kalden JR, Vollmann J. Information and participation in decision-making about treatment: a qualitative study of the perceptions and preferences of patients with rheumatoid arthritis. J Med Ethics. 2008 Nov;34(11):775-9. doi: 10.1136/jme.2007.023705. PMID 18974408
- [Background] Mattukat K, Boehm P, Raberger K, Schaefer C, Keyszer G, Mau W. How Much Information and Participation Do Patients with Inflammatory Rheumatic Diseases Prefer in Interaction with Physicians? Results of a Participatory Research Project. Patient Prefer Adherence. 2019 Dec 17;13:2145-2158. doi: 10.2147/PPA.S209346. eCollection 2019. PMID 31908422
- [Background] Bloem S, Stalpers J, Groenland EAG, van Montfort K, van Raaij WF, de Rooij K. Segmentation of health-care consumers: psychological determinants of subjective health and other person-related variables. BMC Health Serv Res. 2020 Aug 8;20(1):726. doi: 10.1186/s12913-020-05560-4. PMID 32771005
- [Background] Lee YH, Song GG. Relative efficacy and safety of tofacitinib, baricitinib, upadacitinib, and filgotinib in comparison to adalimumab in patients with active rheumatoid arthritis. Z Rheumatol. 2020 Oct;79(8):785-796. doi: 10.1007/s00393-020-00750-1. PMID 32055928